CLINICAL TRIAL: NCT06172790
Title: Investigation of the Effects of the Otago Exercise Program in Adults With Pulmonary Arterial Hypertension Associated With Congenital Heart Disease
Brief Title: The Effects of the Otago Exercise Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cansu Varol, Principal Investigator, Physiotherapist MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-CV-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Arterial Hypertension; Heart Defects, Congenital
Keywords: Otago Exercise Program; Functional Exercise Capacity; Blood Lactate Levels; Quality of Life
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Two groups: training group and control group.
Who Masked: Outcomes Assessor
Masking Description: Our study was conducted as single (assessor) blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The training group will undergo the Otago Exercise Program (OEP) in a hospital setting, supervised by a physiotherapist, with sessions lasting 60 minutes each, three days a week for a duration of 8 weeks.
  Following the initial assessment, a patient education session will be conducted to provide information about the pathophysiology of the disease and the benefits of physical activity.
  Interventions: Other: Training
- Control Group (No Intervention): Any intervention will not be performed. After the initial assessment, a patient education session will be conducted to provide information on the pathophysiology of the disease and the benefits of physical activity.

INTERVENTIONS:
Other: Training — A protocol has been established for the progression of the strengthening and balance training components of the Otago Exercise Program, increasing every two weeks in a four-stage manner. The exercise intensity will be gradually increased based on patient tolerance, ensuring that the perceived difficulty level remains in the range of 4-6 on the Borg dyspnea scale throughout the 8-week period. Supervised walking training is planned to be conducted on a treadmill to ensure standardization. The initial treadmill walking speed for patients will be determined based on the submaximal walking speed in the 6-minute walking test. The progression of the walking program will be carried out every two weeks, similar to the other exercise components of the program, with a 10% increase in walking speed each time.
  Arms: Training Group

SUMMARY:
The objective of this experimental study is to conduct a comparative evaluation of the effects of a supervised Otago Exercise Program (OEP) functional exercise capacity, blood lactate levels, dyspnea, fatigue, peripheral muscle strength, functional mobility, balance performance, quality of life, sleep status, and comorbidities in adults with pulmonary arterial hypertension (PAH) associated with congenital heart disease (CHD), as compared to a control group.

The primary questions driving our study are:

* Does the Otago Exercise Program contribute to an increase in functional capacity?
* Does the Otago Exercise Program have positive effects on blood lactate levels, dyspnea, fatigue, peripheral muscle strength, functional mobility, balance performance, quality of life, sleep status, and comorbidities?

The study participants will be randomly allocated into two groups (n = 50) using a randomized controlled design. The training group (n = 25) will undergo the Otago exercise program, supervised by a physiotherapist, conducted three days a week within a hospital setting for an 8-week intervention period. Following the initial assessment, a patient education session will be administered for the control group (n = 25) and all participants, providing information on disease pathophysiology and the benefits of physical activity. Evaluations will be conducted at baseline and post the 8-week intervention period.

Our research project is designed to investigate the effectiveness of the supervised OEP in adults with CHD associated with PAH. Researchers will compare the training and control groups to determine the effects on functional capacity, blood lactate levels, dyspnea, fatigue, peripheral muscle strength, functional mobility, balance performance, quality of life, sleep status, and comorbidities.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is characterized by a mean pulmonary artery pressure exceeding 20 mmHg, as measured during heart catheterization. In patients with PH, a pulmonary artery wedge pressure of <15 mmHg and a pulmonary vascular resistance of >2 Wood Units indicate the presence of pre-capillary pulmonary hypertension (PubMed ID: 36017548). The current clinical classification for pulmonary arterial hypertension (PAH) associated with congenital heart disease (CHD) comprises four subgroups: Eisenmenger syndrome, left-to-right shunts, coincidental or small defects, and postoperative/closed defects (PubMed ID: 30545968). Prognosis varies based on the type and size of the congenital heart defect, the timing of PAH development, and the response to treatment (PubMed ID:33541620). Adults with PAH associated with CHD exhibit symptoms of dyspnea, cyanosis, chest pain, syncope-presyncope, hemoptysis, decreased exercise capacity, and muscle fatigue (PubMed ID: 34211699). A reduction in exercise capacity is the primary clinical feature of PAH (PubMed ID: 25880178). Compared to other CHD patients, in adults with CHD associated with PAH experience lower exercise tolerance, more severe symptoms, and lower survival rates (PubMed ID: 25896865, 17164490, 21777753). ). The decrease in exercise capacity is linked to the risk of hospitalization or mortality, and exercise intolerance is frequent even in asymptomatic cases (PubMed ID: 16061735). While the benefits of physical activity and exercise in managing chronic diseases are well-established, the therapeutic role of exercise for the CHD-associated PAH population has not been sufficiently investigated (PubMed ID: 32201288). The impact of advanced medical treatment on exercise capacity and quality of life seems to be very limited for this population. Therefore, it is emphasized that additional treatment approaches aimed at improving exercise capacity and quality of life may be necessary for this patient group (PubMed ID: 23041100).

One of the significant symptoms observed in patients with PH is muscle fatigue. In these individuals, adenosine triphosphate is anaerobically produced at lower workloads, leading to early lactic acidosis (PubMed ID: 7856531, 11468205). These changes occur in peripheral muscles may cause to exercise limitation (PubMed ID: 27192047). Elevated lactate levels are associated with anaerobic exercise, this may potentially induced by high pulmonary artery pressure during exercise or deconditioning (PubMed ID: 30464443). Blood lactate concentration stands out as one of the frequently assessed parameters in both clinical exercise testing and performance evaluations of athletes (PubMed ID:19885119). The decrease in physical function has been demonstrated to correlate with a decline in emotional well-being and overall quality of life (PubMed ID: 33660435). Furthermore, a study revealed that maximal isometric forearm muscle strength, assessed with a handgrip in PAH patients, was significantly lower than in their healthy counterparts (PubMed ID: 17689235). Another study comparing PAH patients with healthy individuals reported preserved static balance performance but noted a decrease in dynamic balance performance and balance confidence (PubMed ID: 29251653). In a study conducted by Blok et al., utilizing the Short-form 36 Questionnaire to assess quality of life, it was underscored that the decrease in quality of life serves as a determinant of late-term mortality in patients with CHD-related PAH (PubMed ID: 25911012).

In the guidelines published by the European Society of Cardiology, emphasis is placed on the importance of regular exercise for adults with CHD and CHD associated with PAH. The guidelines encourage patients to engage in regular exercise, receive personalized exercise prescriptions, and maintain an active lifestyle. Structured regular exercise is deemed a safe and effective treatment for most patients with CHD (PubMed ID: 32860412, 32860028). ). In the literature, exercise training programs have been implemented for adults with CHD associated with PAH, both in home- and hospital-based settings, with or without supervision (PubMed ID: 23041100, 20136857). There are studies in the literature have explored the effects of aerobic and resistance training, as well as respiratory muscle training (PubMed ID: 23041100, 19604588, 20136857).

The Otago Exercise Program (OEP) is an evidence-based multimodal exercise regimen developed by Campbell and the Otago Medical School of New Zealand in 1997 (PubMed ID: 9366737). Widely utilized during rehabilitation and the postoperative recovery period, the OEP has been studied in various conditions such as osteoarthritis, rheumatoid arthritis, knee prosthesis postoperative rehabilitation, Parkinson's and Alzheimer's disease, stroke, visual impairment, depression, dementia, and cognitive impairment. Recognized as a safe protocol, it is predominantly applied in the literature as a home exercise program for the geriatric population residing in the community. Moreover, recent studies have adapted it to Kinect technologies, presenting virtual exercises, and implemented it as a telehealth service with a home-based exercise program during the Covid-19 pandemic period (PubMed ID: 31118594, 34289524, 19607686, 20458104, 33225343, 28827207, 29958232, 36339194).

Physical activity recommendations for adults with CHD associated with PAH often advise against vigorous intensity exercise in numerous guidelines. The Otago Exercise Program, chosen as an evidence-based multimodal exercise regimen to establish a safe exercise prescription, aligns with literature recommendations. This upcoming study, focusing in adults with CHD associated with PAH a population known for low exercise capacity with recommendations for further research aims to formulate exercise training strategies beneficial for patients.

Our study will be the first investigation examining the effects of the Otago Exercise Program implemented under physiotherapist supervision. With this study to be conducted in adults with congenital heart disease associated pulmonary arterial hypertension, who are reported to have low exercise capacity and further research is recommended, the aim is to develop exercise training strategies that will benefit patients.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically and hemodynamically stable.
* Resting mean pulmonary artery pressure measured with left heart catheterization to be 20 mmHg or higher.
* Being 18 years of age or older.
* Being classified as World Health Organization-functional class II and III.
* Being under optimized advanced medical treatment for PAH for at least 2 months before entering the study.
* No changes in pulmonary arterial hypertension medical treatment for at least 6 months before entering the study.

Exclusion Criteria:

* The coexistence of Down syndrome.
* Group 1 PAH patients with another etiology.
* Changes in PAH medical treatment during follow-up.
* Acute decompensated heart failure.
* Unstable angina pectoris.
* Recent thoracic or abdominal surgeries.
* Using immunosuppressive drugs due to organ or tissue transplantation.
* Heavy neurological disorders causing autonomic dysfunction.
* The presence of cognitive impairment preventing communication.
* Recent syncope, fractures, osteoporosis, presence of tumors, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The Six-Minute Walk Test | Change from Baseline at 8 weeks
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society. Functional exercise capacity will be evaluated with the six-minute walk test. Patients will be walked in a 30-meter-long corridor for 6 minutes and the maximum walking distance will be measured. Before and after the test, heart rate, blood pressure and O2 saturation will be measured with pulse oximetry, and dyspnea and fatigue levels will be determined according to the Modified Borg scale.

SECONDARY OUTCOMES:
Duke Activity Status Index | Change from Baseline at 8 weeks
  The Duke Activity Status Index includes self care, ambulation, household tasks, sexual function and recreational activities. Maximal oxygen consumption values for the cases will be obtained using the formula based on the Duke Activity Status Index result. As a result of scoring, a total score ranging from 0 to 58.2 is obtained. Higher scores indicate higher functional capacity.
Blood Lactate Levels | Change from Baseline at 8 weeks
  Before, immediately after, and 5 minutes after the six-minute walk test, three measurements will be taken using a portable lactate measurement device.
Modified Borg Scale | Change from Baseline at 8 weeks
  The Modified Borg Scale is used to determine the level of breathlessness and fatigue at rest and during exertion. Before and after the six-minute walk test, the levels of dyspnea and fatigue will be evaluated using 'Modified Borg Dyspnea' and 'Modified Borg Fatigue.' It consists of 10 items that define the intensity of breathlessness and fatigue on a scale ranging from 0 (none) to 10 (very severe). A rating of "0" means you feel no breathlessness and fatigue. From 0 to 10, symptoms worsen.
Peripheral Muscle Strength Assessment | Change from Baseline at 8 weeks
  Hand grip strength will be assessed with a hydraulic hand dynamometer while the patient is in a seated position, following the guidelines of the American Society of Hand Therapists. The highest scores within the measurements will be recorded as hand grip strength in kilograms.
30-Second Sit-to-Stand Test | Change from Baseline at 8 weeks
  Functional mobility and balance performances are assessed. The patient will be instructed to sit in the middle of a standard chair with feet touching the ground and arms crossed on the chest. The test begins with the 'start' command, and the patient is asked to perform as many full stands as possible within a 30-second period. The number of full stands completed by the patient during the 30-second interval is recorded.
Timed Up and Go Test | Change from Baseline at 8 weeks
  A standard chair is used for the test. Initially, the patient is asked to sit on the chair with support. Subsequently, the patient is instructed to stand up, walk with regular steps over a predetermined distance of 3 meters, turn around at the end of the 3 meters, and return to sit back on the chair. The time taken by the patient to complete the test is recorded. A shorter duration indicates better performance. Functional mobility and balance performances are assessed.
Four-Stage Balance Test | Change from Baseline at 8 weeks
  The balance is assessed for 10 seconds in four different positions and the total time is summed. Stages are passed if the patient can hold the stance for 10 seconds. An inability to maintain tandem stance for 10 seconds with eyes open is associated with higher risk of falling. For scoring purposes, a score of 1 (success) is recorded for each test position if the participant was able to complete the task for 10 seconds; If the task is not completed within 10 seconds, a score of 0 (failure) is recorded. Scores (range: 0-4) are sum across the four test conditions, with higher values indicating better balance.
The emPHasis-10 Questionnaire | Change from Baseline at 8 weeks
  The emPHasis-10 questionnaire will be used to measure quality of life. The emPHasis-10, as a single-dimensional, easily applicable, short questionnaire, consists of 10 simple questions addressing concerns related to fatigue, dyspnea, lack of energy, social limitations, and the impact on family members. Each question is scored on a Likert scale of 0-5. The total score ranges from 0 to 50, with a higher score indicating a deterioration in quality of life due to pulmonary hypertension symptoms.
Pittsburgh Sleep Quality Index | Change from Baseline at 8 weeks
  The Pittsburgh Sleep Quality Index is a 10-item self-report questionnaire that is designed to measure sleep quality in clinical populations, and assess usual sleep habits during the past one-month. This scale generates seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Items 1-4 inquire about the amount of sleep and responses are recorded in free-text boxes. Items 5-10 inquire about specific sleep behaviors and quality, which are rated on 4-point scale. Finally, the scores for each component are summed to get a total score, also termed the global score (range: 0 to 21). A global sum of "5"or greater indicates a "poor" sleeper.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof, Study Director — Istanbul University - Cerrahpasa (IUC) Cardiology Institute; Mehmet Serdar Kucukoglu, Prof, Study Chair — Istanbul University - Cerrahpasa (IUC) Cardiology Institute
Locations (1):
- Istanbul University - Cerrahpasa (IUC) Cardiology Institute, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Heart J. 2022 Oct 11;43(38):3618-3731. doi: 10.1093/eurheartj/ehac237. No abstract available. PMID 36017548
- [Background] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Background] Rosenzweig EB, Krishnan U. Congenital Heart Disease-Associated Pulmonary Hypertension. Clin Chest Med. 2021 Mar;42(1):9-18. doi: 10.1016/j.ccm.2020.11.005. Epub 2021 Jan 12. PMID 33541620
- [Background] Kucukoglu SM, Kaymaz C, Alehan D, Kula S, Akcevin A, Celiker A, Cicek SM, Tokgozoglu LS, Kentli S; THALES Registry Investigators. Pulmonary arterial hypertension associated with congenital heart disease: lessons learnt from the large Turkish Nationwide Registry (THALES). Pulm Circ. 2021 Jun 18;11(3):20458940211024206. doi: 10.1177/20458940211024206. eCollection 2021 Jul-Sep. PMID 34211699
- [Background] Demir R, Kucukoglu MS. Six-minute walk test in pulmonary arterial hypertension. Anatol J Cardiol. 2015 Mar;15(3):249-54. doi: 10.5152/akd.2015.5834. PMID 25880178
- [Background] Bhatt AB, Foster E, Kuehl K, Alpert J, Brabeck S, Crumb S, Davidson WR Jr, Earing MG, Ghoshhajra BB, Karamlou T, Mital S, Ting J, Tseng ZH; American Heart Association Council on Clinical Cardiology. Congenital heart disease in the older adult: a scientific statement from the American Heart Association. Circulation. 2015 May 26;131(21):1884-931. doi: 10.1161/CIR.0000000000000204. Epub 2015 Apr 20. No abstract available. PMID 25896865
- [Background] Engelfriet PM, Duffels MG, Moller T, Boersma E, Tijssen JG, Thaulow E, Gatzoulis MA, Mulder BJ. Pulmonary arterial hypertension in adults born with a heart septal defect: the Euro Heart Survey on adult congenital heart disease. Heart. 2007 Jun;93(6):682-7. doi: 10.1136/hrt.2006.098848. Epub 2006 Dec 12. PMID 17164490
- [Background] Lowe BS, Therrien J, Ionescu-Ittu R, Pilote L, Martucci G, Marelli AJ. Diagnosis of pulmonary hypertension in the congenital heart disease adult population impact on outcomes. J Am Coll Cardiol. 2011 Jul 26;58(5):538-46. doi: 10.1016/j.jacc.2011.03.033. PMID 21777753
- [Background] Diller GP, Dimopoulos K, Okonko D, Li W, Babu-Narayan SV, Broberg CS, Johansson B, Bouzas B, Mullen MJ, Poole-Wilson PA, Francis DP, Gatzoulis MA. Exercise intolerance in adult congenital heart disease: comparative severity, correlates, and prognostic implication. Circulation. 2005 Aug 9;112(6):828-35. doi: 10.1161/CIRCULATIONAHA.104.529800. Epub 2005 Aug 1. PMID 16061735
- [Background] Tran D, Maiorana A, Ayer J, Lubans DR, Davis GM, Celermajer DS, d'Udekem Y, Cordina R. Recommendations for exercise in adolescents and adults with congenital heart disease. Prog Cardiovasc Dis. 2020 May-Jun;63(3):350-366. doi: 10.1016/j.pcad.2020.03.002. Epub 2020 Mar 19. PMID 32201288
- [Background] Becker-Grunig T, Klose H, Ehlken N, Lichtblau M, Nagel C, Fischer C, Gorenflo M, Tiede H, Schranz D, Hager A, Kaemmerer H, Miera O, Ulrich S, Speich R, Uiker S, Grunig E. Efficacy of exercise training in pulmonary arterial hypertension associated with congenital heart disease. Int J Cardiol. 2013 Sep 20;168(1):375-81. doi: 10.1016/j.ijcard.2012.09.036. Epub 2012 Oct 5. PMID 23041100
- [Background] Nootens M, Wolfkiel CJ, Chomka EV, Rich S. Understanding right and left ventricular systolic function and interactions at rest and with exercise in primary pulmonary hypertension. Am J Cardiol. 1995 Feb 15;75(5):374-7. doi: 10.1016/s0002-9149(99)80557-8. PMID 7856531
- [Background] Sun XG, Hansen JE, Oudiz RJ, Wasserman K. Exercise pathophysiology in patients with primary pulmonary hypertension. Circulation. 2001 Jul 24;104(4):429-35. doi: 10.1161/hc2901.093198. PMID 11468205
- [Background] Babu AS, Arena R, Myers J, Padmakumar R, Maiya AG, Cahalin LP, Waxman AB, Lavie CJ. Exercise intolerance in pulmonary hypertension: mechanism, evaluation and clinical implications. Expert Rev Respir Med. 2016 Sep;10(9):979-90. doi: 10.1080/17476348.2016.1191353. Epub 2016 Jun 10. PMID 27192047
- [Background] Skjorten I, Hilde JM, Melsom MN, Hisdal J, Hansteen V, Steine K, Humerfelt S. Exercise capacity in COPD patients with exercise-induced pulmonary hypertension. Int J Chron Obstruct Pulmon Dis. 2018 Oct 31;13:3599-3610. doi: 10.2147/COPD.S161175. eCollection 2018. PMID 30464443
- [Background] Goodwin ML, Harris JE, Hernandez A, Gladden LB. Blood lactate measurements and analysis during exercise: a guide for clinicians. J Diabetes Sci Technol. 2007 Jul;1(4):558-69. doi: 10.1177/193229680700100414. PMID 19885119
- [Background] Constantine A, Condliffe R, Clift P, Tulloh R, Dimopoulos K; CHAMPION Steering Committee. Palliative care in pulmonary hypertension associated with congenital heart disease: systematic review and expert opinion. ESC Heart Fail. 2021 Jun;8(3):1901-1914. doi: 10.1002/ehf2.13263. Epub 2021 Mar 3. PMID 33660435
- [Background] Bauer R, Dehnert C, Schoene P, Filusch A, Bartsch P, Borst MM, Katus HA, Meyer FJ. Skeletal muscle dysfunction in patients with idiopathic pulmonary arterial hypertension. Respir Med. 2007 Nov;101(11):2366-9. doi: 10.1016/j.rmed.2007.06.014. Epub 2007 Aug 6. PMID 17689235
- [Background] Ozcan Kahraman B, Ozsoy I, Savci S, Acar S, Ozpelit E, Sevinc C, Akdeniz B. Static and Dynamic Balance Performance and Balance Confidence in Individuals With and Without Pulmonary Arterial Hypertension. J Cardiopulm Rehabil Prev. 2018 Jul;38(4):259-263. doi: 10.1097/HCR.0000000000000299. PMID 29251653
- [Background] Blok IM, van Riel AC, Schuuring MJ, Duffels MG, Vis JC, van Dijk AP, Hoendermis ES, Mulder BJ, Bouma BJ. Decrease in quality of life predicts mortality in adult patients with pulmonary arterial hypertension due to congenital heart disease. Neth Heart J. 2015 May;23(5):278-84. doi: 10.1007/s12471-015-0666-9. PMID 25911012
- [Background] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412
- [Background] Martinez-Quintana E, Miranda-Calderin G, Ugarte-Lopetegui A, Rodriguez-Gonzalez F. Rehabilitation program in adult congenital heart disease patients with pulmonary hypertension. Congenit Heart Dis. 2010 Jan-Feb;5(1):44-50. doi: 10.1111/j.1747-0803.2009.00370.x. PMID 20136857
- [Background] Giannakoulas G, Dimopoulos K. Exercise training in congenital heart disease: should we follow the heart failure paradigm? Int J Cardiol. 2010 Jan 21;138(2):109-11. doi: 10.1016/j.ijcard.2009.06.024. Epub 2009 Jul 14. PMID 19604588
- [Background] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Background] Cederbom S, Arkkukangas M. Impact of the fall prevention Otago Exercise Programme on pain among community-dwelling older adults: a short- and long-term follow-up study. Clin Interv Aging. 2019 Apr 26;14:721-726. doi: 10.2147/CIA.S200188. eCollection 2019. PMID 31118594
- [Background] Chen X, Zhao L, Liu Y, Zhou Z, Zhang H, Wei D, Chen J, Li Y, Ou J, Huang J, Yang X, Ma C. Otago exercise programme for physical function and mental health among older adults with cognitive frailty during COVID-19: A randomised controlled trial. J Clin Nurs. 2025 Dec;34(12):5130-5143. doi: 10.1111/jocn.15964. Epub 2021 Jul 21. PMID 34289524
- [Background] Hill KD, LoGiudice D, Lautenschlager NT, Said CM, Dodd KJ, Suttanon P. Effectiveness of balance training exercise in people with mild to moderate severity Alzheimer's disease: protocol for a randomised trial. BMC Geriatr. 2009 Jul 16;9:29. doi: 10.1186/1471-2318-9-29. PMID 19607686
- [Background] Kerse N, Hayman KJ, Moyes SA, Peri K, Robinson E, Dowell A, Kolt GS, Elley CR, Hatcher S, Kiata L, Wiles J, Keeling S, Parsons J, Arroll B. Home-based activity program for older people with depressive symptoms: DeLLITE--a randomized controlled trial. Ann Fam Med. 2010 May-Jun;8(3):214-23. doi: 10.1370/afm.1093. PMID 20458104
- [Background] Liu-Ambrose T, Davis JC, Falck RS, Best JR, Dao E, Vesely K, Ghag C, Rosano C, Hsu CL, Dian L, Cook W, Madden KM, Khan KM. Exercise, Processing Speed, and Subsequent Falls: A Secondary Analysis of a 12-Month Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2021 Mar 31;76(4):675-682. doi: 10.1093/gerona/glaa239. PMID 33225343
- [Background] Mat S, Ng CT, Tan PJ, Ramli N, Fadzli F, Rozalli FI, Mazlan M, Hill KD, Tan MP. Effect of Modified Otago Exercises on Postural Balance, Fear of Falling, and Fall Risk in Older Fallers With Knee Osteoarthritis and Impaired Gait and Balance: A Secondary Analysis. PM R. 2018 Mar;10(3):254-262. doi: 10.1016/j.pmrj.2017.08.405. Epub 2017 Aug 18. PMID 28827207
- [Background] Shubert TE, Chokshi A, Mendes VM, Grier S, Buchanan H, Basnett J, Smith ML. Stand Tall-A Virtual Translation of the Otago Exercise Program. J Geriatr Phys Ther. 2020 Jul/Sep;43(3):120-127. doi: 10.1519/JPT.0000000000000203. PMID 29958232
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194
- [Background] Baumgartner H, De Backer J, Babu-Narayan SV, Budts W, Chessa M, Diller GP, Lung B, Kluin J, Lang IM, Meijboom F, Moons P, Mulder BJM, Oechslin E, Roos-Hesselink JW, Schwerzmann M, Sondergaard L, Zeppenfeld K; ESC Scientific Document Group. 2020 ESC Guidelines for the management of adult congenital heart disease. Eur Heart J. 2021 Feb 11;42(6):563-645. doi: 10.1093/eurheartj/ehaa554. No abstract available. PMID 32860028